CLINICAL TRIAL: NCT07273266
Title: The Effect of Routine Versus Random Pacifier Administration Methods on Feeding Maturity in Preterm Infants
Brief Title: Feeding Maturity in Preterm Infants
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Zehra Kan Onturk, Assoc. Prof., Acibadem University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ATADEK-2024/19
Record Dates: First submitted 2025-11-25; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Preterm; Feeding; Non Nutritive Sucking
Keywords: preterm; feeding; non nutritive sucking; feeding maturation
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine NNS (Experimental): Newborns who receive routine 5-minute pacifier use before each feeding will constitute the intervention group.
  Interventions: Device: Routine NNS
- Control group (Random NNS) (Other): Newborns who are given a pacifier for 30 minutes at random times throughout the day, independent of feeding and based on the infant's cues, will constitute the control group.
  Interventions: Device: Random NNS

INTERVENTIONS:
Device: Routine NNS — The content, volume, and method of feeding are determined by the physician. A pacifier is provided for 5 minutes before each feeding. Procedures are carried out in accordance with the "Newborn Nursing Protocols," based on the infant's feeding method.
  Feeding maturity is assessed once a week using a feeding monitor.
  Arms: Routine NNS
Device: Random NNS — The content, volume, and method of feeding are determined by the physician. The infant is given a pacifier for 30 minutes at random times during the day, independent of feeding.
  Procedures are carried out in accordance with the "Newborn Nursing Protocols," based on the infant's feeding method.
  Feeding maturity is assessed once a week using a feeding monitor.
  Arms: Control group (Random NNS)

SUMMARY:
The aim of this study is to evaluate the effect of two pacifier-use strategies-routine 5-minute pacifier use prior to each feeding versus random 30-minute pacifier use at any time of day, independent of feeding-on feeding maturity in preterm infants. The hypotheses of the study are as follows: H1: The routine use of a pacifier prior to feeding has a positive effect on feeding maturity in preterm infants.

H2: The routine use of a pacifier prior to feeding has a positive effect on discharge weight in preterm infants.

H3: The routine use of a pacifier prior to feeding has a positive effect on the length of hospital stay in preterm infants.

H4: The routine use of a pacifier prior to feeding has a positive effect on the gestational age at discharge in preterm infants.

DETAILED DESCRIPTION:
Developing safe and effective feeding skills in preterm infants is a highly complex process. To achieve feeding maturity, preterm infants must establish oropharyngeal anatomical integrity, adequate neurological function, and full coordination of sucking, swallowing, and breathing. Due to this immaturity, they frequently experience oral feeding difficulties such as low oral-motor tone, poor suck-swallow-breath coordination, sleepiness, gastrointestinal dysmotility, immature sucking pressure, and an inability to maintain stable physiological parameters during feeding. Effective oral feeding is crucial for optimal growth, safe discharge, and the prevention of aspiration and long-term respiratory or neurological complications.

For this reason, preterm infants require support until they develop the necessary skills for oral feeding and successfully transition from orogastric tube feeding to total oral intake. During this transition period, early oral stimulation methods help promote oral development and self-regulation. Among these supportive and complementary strategies, non-nutritive sucking (NNS) facilitates the progression toward oral feeding. Evidence indicates that infants who receive NNS transition to full oral feeding more quickly, demonstrate better feeding performance, achieve more organized sucking behavior, experience improved digestion, and remain more active during feeds.

Although studies emphasize the benefits of NNS, research examining how the frequency, duration, or timing of NNS influences feeding maturity remains limited.

ELIGIBILITY:
Inclusion Criteria:

* Preterm
* who are clinically stable, and
* who are within the first day of initiating enteral feeding.

Exclusion Criteria:

* Newborns who have a contraindication to pacifier use
* have comorbid medical conditions
* who are intubated
* have congenital anomalies

Ages: 0 Days to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 62 (Estimated)
Dates: Start 2025-03-04 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Feeding maturity | From the start of oral feeding until hospital discharge; assessed weekly for up to 6 weeks. The change in these time intervals will be assessed.
  Feeding maturity will be evaluated using a feeding monitor, assessing key swallowing and respiratory coordination parameters, including the number and duration of rhythmic swallows, rest periods, swallow-respiration patterns, and total milk volume consumed.

SECONDARY OUTCOMES:
Change in Body Weight | From initiation of total oral feeding to hospital discharge (average 5 weeks)
  Participant's body weight will be assessed at initiation of total oral feeding and at hospital discharge.
Length of Hospital Stay | From baseline to discharge (average 15 weeks)
  The time from date of hospitalization until the date of discharge.
Age at discharge | At first discharge home, on average 37 weeks postmenstrual age
  Postmenstrual age (weeks) of the infant at the time of hospital discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Serdar Beken, Principal Investigator — Acibadem University
Locations (1):
- Acıbadem University, Istanbul, Ataşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Foster JP, Psaila K, Patterson T. Non-nutritive sucking for increasing physiologic stability and nutrition in preterm infants. Cochrane Database Syst Rev. 2016 Oct 4;10(10):CD001071. doi: 10.1002/14651858.CD001071.pub3. PMID 27699765
- [Background] Kaya V, Aytekin A. Effects of pacifier use on transition to full breastfeeding and sucking skills in preterm infants: a randomised controlled trial. J Clin Nurs. 2017 Jul;26(13-14):2055-2063. doi: 10.1111/jocn.13617. Epub 2017 Mar 21. PMID 27754572
- [Background] Ecevit A, Erdogan B, Anuk Ince D, Aksu M, Unal S, Turan O, Saracoglu A, Tarcan A. Determination of oral feeding skills in late preterm, early term, and full-term infants using the neonatal oral feeding monitor (NeoSAFE). Ital J Pediatr. 2025 Feb 7;51(1):38. doi: 10.1186/s13052-025-01867-2. PMID 39920842
- [Background] Munoz-Gomez E, Ingles M, Molla-Casanova S, Sempere-Rubio N, Serra-Ano P, Aguilar-Rodriguez M. Effects of an Oral Stimulation Program on Feeding Outcomes in Preterm Infants: A Systematic Review and Meta-Analysis. Phys Occup Ther Pediatr. 2024;44(1):110-127. doi: 10.1080/01942638.2023.2212767. Epub 2023 May 18. PMID 37203152
- [Background] Zhao S, Jiang H, Miao Y, Liu W, Li Y, Zhang Y, Wang A, Cui X. Effects of implementing non-nutritive sucking on oral feeding progression and outcomes in preterm infants: A systematic review and meta-analysis. PLoS One. 2024 Apr 16;19(4):e0302267. doi: 10.1371/journal.pone.0302267. eCollection 2024. PMID 38626172